CLINICAL TRIAL: NCT00093067
Title: A Phase 3, Multicenter, Randomized, Open-Label, Comparative Study to Assess the Safety and Efficacy of Daptomycin Compared to Conventional Therapy In the Treatment of Subjects With Infective Endocarditis or Bacteremia Due to Staph Aureus
Brief Title: Daptomycin in the Treatment of Subjects With Infective Endocarditis or Bacteremia Due to S. Aureus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3009-007; DAP-IE-01-02 (Other: Cubist)
Record Dates: First submitted 2004-09-30; First posted 2004-10-01 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Bacterial Endocarditis; Bacteremia
Keywords: Gram-positive bacterial infections; Staph Aureus; endocarditis; bacteremia; Cubist
MeSH Terms: conditions — Endocarditis, Bacterial; Bacteremia; Gram-Positive Bacterial Infections; Staphylococcal Infections; Endocarditis | interventions — Daptomycin

INTERVENTIONS:
Drug: daptomycin

SUMMARY:
The purpose of this study is to compare the safety and efficacy of daptomycin, an antibiotic, to standard therapy in subjects who have infective endocarditis or bacteremia due to Staphylococcus aureus (S. aureus).

DETAILED DESCRIPTION:
Even with prompt treatment, Staphylococcus aureus Infective Endocarditis (IE) continues to be associated with significant morbidity and mortality indicating a need for new therapeutic approaches. In vitro, daptomycin is rapidly bactericidal, with concentration-dependent killing, and MIC90 of 0.5 microgram/ml for S. aureus; in clinical studies, daptomycin appears to be well tolerated and can be administered once every 24 hours by i.v. infusion. These characteristics suggest it should be clinically and microbiologically effective in the treatment of serious S. aureus infections, including IE and bacteremia

Comparison: standard of care (Vancomycin or Semi-synthetic Penicillin with adjunct gentamicin)

ELIGIBILITY:
Inclusion Criteria:

* Documented S. aureus bacteremia within 2 calendar days of the first dose of study medication

Exclusion Criteria:

* Subjects with a creatinine clearance of less than 30 ml/min
* Subjects with pneumonia
* Pregnant, nursing, or lactating
* Documented history of allergy or intolerance to penicillin or vancomycin
* Subjects with osteomyelitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-03; Primary Completion 2004-11 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
To demonstrate that daptomycin is not inferior to comparator in the treatment of S. aureus bacteremia and IE as assessed by the Independent External Adjudication Committee (IEAC) Outcome at Test of Cure (TOC) in the Intention-to-Treat (ITT) population.

SECONDARY OUTCOMES:
To compare clinical success rates between daptomycin and comparator in the treatment of S. aureus bacteremia and IE as assessed by the IEAC Outcome at End of Treatment (EOT) in the ITT population.
To compare clinical success rates between daptomycin and comparator in the treatment of S. aureus bacteremia and IE as assessed by the IEAC Outcome at EOT and TOC in the Per Protocol (PP) population.
To compare clinical success rates between daptomycin and comparator in the treatment of S. aureus bacteremia and IE as assessed by the IEAC Outcome for each of the diagnoses defined by the IEAC at EOT in the ITT population.
To compare clinical success rates between daptomycin and comparator in the treatment of S. aureus bacteremia and IE as assessed by the IEAC Outcome for each of the diagnoses defined by the Investigator at EOT in the ITT population.
To compare microbiologic eradication rates between daptomycin and comparator.
To demonstrate that survival rates are similar between daptomycin and comparator in the ITT population.
To evaluate the safety of daptomycin as compared to comparator in the safety population.
To assess the pharmacokinetics of daptomycin.
To compare the pharmacoeconomic impact of daptomycin with that of comparator.

REFERENCES:
- [Result] Fowler VG Jr, Boucher HW, Corey GR, Abrutyn E, Karchmer AW, Rupp ME, Levine DP, Chambers HF, Tally FP, Vigliani GA, Cabell CH, Link AS, DeMeyer I, Filler SG, Zervos M, Cook P, Parsonnet J, Bernstein JM, Price CS, Forrest GN, Fatkenheuer G, Gareca M, Rehm SJ, Brodt HR, Tice A, Cosgrove SE; S. aureus Endocarditis and Bacteremia Study Group. Daptomycin versus standard therapy for bacteremia and endocarditis caused by Staphylococcus aureus. N Engl J Med. 2006 Aug 17;355(7):653-65. doi: 10.1056/NEJMoa053783. PMID 16914701
- [Derived] Bhavnani SM, Rubino CM, Ambrose PG, Drusano GL. Daptomycin exposure and the probability of elevations in the creatine phosphokinase level: data from a randomized trial of patients with bacteremia and endocarditis. Clin Infect Dis. 2010 Jun 15;50(12):1568-74. doi: 10.1086/652767. PMID 20462352